CLINICAL TRIAL: NCT02845492
Title: Testing the Effects of Qigong on a Multi-System Neuro-muscular- Immune Model of Vigor in Cancer Survivorship
Brief Title: Evaluating Qigong as a Clinical Intervention for Cancer Survivors' Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Catherine Kerr, Assistant Professor of Family Medicine, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MiriamH
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Fatigue
Keywords: Exercise; Qigong; Mind-Body; Fatigue; Cancer; EEG; HRV
MeSH Terms: conditions — Fatigue; Motor Activity; Neoplasms | interventions — Qigong

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qigong intervention (Experimental): Qigong meditative exercise intervention meets three times a week for 10 weeks. The qigong group (n=30) will meet at the Women's Medicine Collaborative, Miriam Hospital (146 W. River St., Providence, RI) for Qigong classes. The lesson will be taught by a validated Qi Gong master with over forty years of experience and the interventional protocol will be validated. Two and a half hours of weekly outside personal practice will also be required of participants.
  Interventions: Other: Qigong
- CHIP healthy wellness-exercise class (Active Comparator): The Complete Health Improvement Program is a validated set of weekly classes designed to promote gentle exercise and wellness related activities in a supportive group setting led by an experienced trainer.
  Interventions: Other: Complete Health Improvement Program (CHIP)

INTERVENTIONS:
Other: Qigong — Qigong is a mind-body exercise based around gentle exercise and the cultivation of a meditative focus on bodily sensations
  Other Names: Meditative Exercise Therapy
  Arms: Qigong intervention
Other: Complete Health Improvement Program (CHIP) — The CHIP program is a validated weekly wellness and exercise program designed to promote health and wellbeing.
  Other Names: Wellness-Exercise Program
  Arms: CHIP healthy wellness-exercise class

SUMMARY:
This study compares Qigong movement-based meditation exercise with a healthy living exercise-wellness course. There are two primary goals of this research:

1. Evaluate and compare physiological mechanisms underlying the two wellness-exercise interventions with the specific goal of understanding the physiology of Qigong.

   Using a simple noninvasive EEG setup, the study will test some of the same brain mechanisms that have been found in mindfulness meditation.

   The study will also investigate Qigong's effects on stress and heart signals and on inflammation in the immune system. A key hypothesis is that Qigong will show distinctive, stronger effects on brain and heart measures. A related hypothesis is that Qigong will show stronger effects on blood markers of inflammation.
2. Compare effect sizes of the two interventions in decreasing fatigue in order to plan for a larger clinical trial.

DETAILED DESCRIPTION:
Between 20-50% of Cancer Survivors report fatigue following treatment that interferes with their daily life. However, to date no treatment option has been definitively validated as effective for fatigue in survivors. In recent years Mind Body exercises such as yoga, Tai Chi, and Qigong have been shown in small clinical trials to be effective at treating the symptoms of CRF in a wide array of Cancer types. But understanding of basic science mechanisms is poor.

Recent studies of Mindfulness meditation, by the investigators and others, confirm the importance of brain mechanisms related to awareness and attention. This study will assess whether Qigong activates similar physiological processes. The study will also assess (1) whether emotion regulation improves, suggesting that Mindfulness-related processes may partially underlie changes in Qigong as a Mindful exercise (2) whether grip strength improves, suggesting that Qigong activates similar processes to conventional exercise.

As an exploratory question, the study will look at whether brain measures related to awareness are correlated with inflammatory markers called cytokines, suggesting possible neuro-immune interaction that may be relevant for understanding fatigue, vitality and embodied meditative movement therapies such as Qigong, Tai Chi and Yoga.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 18-70 years
* Self-report of fatigue =/> 3/10 on fatigue interference scale
* Have been diagnosed and completed treatment for cancer (with surgery or radiation or chemotherapy)
* no surgery, radiation or chemotherapy received in the past 8 weeks (ongoing treatment with Herceptin [trastuzumab] or other adjuvant therapies is permitted)
* Currently cancer-free
* Have a primary care or other physician
* Ability to understand English
* Willingness to have blood drawn, have an EEG taken and complete questionnaires
* Ability to pass basic validated physical movement tests (e.g.: standing with feet touching for 30 seconds, twist right to left and back, hold arms out to side in air for 15 seconds, lift arms over head, moving from standing position to seated position on the floor) to verify safety for Qigong practice.

Exclusion Criteria:

* History or current diagnosis of medical or psychiatric disorder that would interfere with ability to participate in wellness classes or in scientific assessment sessions (e.g., rheumatoid arthritis, diabetes, major psychiatric disorder, connective tissue disorder)
* Body Mass Index (BMI) > 31
* Active alcohol or drug abuse
* Tobacco use
* Pregnancy
* Regular daily use of anti-inflammatory drugs, including non-steroidal anti-inflammatory drugs, (does not apply to common use of daily "baby aspirin" as daily prophylactic cardiovascular treatment)
* Resting systolic blood pressure of less than 90 or greater than 160 and resting diastolic blood pressure of greater than 110.
* Ingestion of caffeine or cocoa products less than two hours from data collection
* Contraindication to regular physical activity participation
* Already engaging in >60 min of vigorous physical activity per week for the prior month
* Weekly practice of yoga, Tai Chi, Qigong, or meditation since the diagnosis of cancer
* Peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory Questionnaire | Change from baseline to 10 weeks
  Questions about daily experience of fatigue

SECONDARY OUTCOMES:
EEG meditative brain measures, | at baseline and at 10 weeks
  Acquired using a non-invasive EEG cap that sits on the scalp
Self-reported Vitality (a component of the Medical Outcomes Short-Form 36) | at baseline and 10 weeks
Heart Rate Variability (HRV) | at baseline and 10 weeks
  Acquired using an EKG
Inflammatory cytokines | at baseline and 10 weeks
  Cytokine measures: Il-1, Il-6, Il-10, tnf-alpha

OTHER OUTCOMES:
Difficulties in emotion regulation self-report scale (DERS) | at baseline and 10 weeks
  Questions about emotions and emotion regulation
Handgrip strength | at baseline and 10 weeks
  Uses dynamometer to assess handgrip strength

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Kerr, PhD, Principal Investigator — Women's Medicine Collaborative, Miriam Hospital
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be archived with with computer scripts into a package. These packages will be available to any investigator who requests them.

REFERENCES:
- [Background] Kerr CE, Sacchet MD, Lazar SW, Moore CI, Jones SR. Mindfulness starts with the body: somatosensory attention and top-down modulation of cortical alpha rhythms in mindfulness meditation. Front Hum Neurosci. 2013 Feb 13;7:12. doi: 10.3389/fnhum.2013.00012. eCollection 2013. PMID 23408771
- [Background] Schmalzl L, Kerr CE. Editorial: Neural Mechanisms Underlying Movement-Based Embodied Contemplative Practices. Front Hum Neurosci. 2016 Apr 26;10:169. doi: 10.3389/fnhum.2016.00169. eCollection 2016. No abstract available. PMID 27199700